CLINICAL TRIAL: NCT06864936
Title: Exploration of Novel Imaging Biomarkers on OCT for Ublituximab Treatment Response in Multiple Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: TG Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Daniel Harrison, Principal Investigator, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00113916
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis (MS) - Relapsing-remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — ublituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ublituximab (Active Comparator): Subjects recently prescribed ublituximab will undergo a specialized OCT at Enrollment, Month 6 and Month 12 as well as other neurologic assessments typically used in MS clinical trials such as EDSS, MSFC and SDMT
  Interventions: Drug: Ublituximab
- Other Disease Modifying Therapy (Active Comparator): People on stable doses of non-B-cell depleting multiple sclerosis disease modifying therapies will undergo the specialized OCT scan at baseline, 6 months, and 12 months.
  Interventions: Other: Other disease modifying therapies

INTERVENTIONS:
Drug: Ublituximab — ublituximab
  Arms: Ublituximab
Other: Other disease modifying therapies — Other disease modifying therapies for MS (not ublituximab)
  Arms: Other Disease Modifying Therapy

SUMMARY:
The purpose of the research study is to explore new retinal imaging biomarkers of immune cell activity in MS during use of ublituximab (Briumvi) treatment. A biomarker is a biological molecule found in blood, other body fluids, or tissues that is a sign of a normal or abnormal process, or of a condition or disease. A biomarker may be used to see how well the body responds to a treatment for a disease or condition. This study will evaluate the efficacy of ublituximab to modulate MS pathology in a new manner. In order to assess this new biomarker, a specialized optical coherence tomography (OCT) scan will be performed at enrollment into the study and at 2 other timepoints throughout the study.

Subjects asked to take part in this study should have been diagnosed with relapsing multiple sclerosis (MS) and have recently been advised to start the medication ublituximab (Briumvi) or are currently on another medication for the treatment of their MS.

We plan to enroll 30 patients into this study. Fifteen (15) patients with Relapsing Remitting Multiple Sclerosis (RRMS) who are being initiated on B-cell depletion therapy by their treating physician at the University of Maryland Center for MS Treatment and Research will be offered enrollment into this study. Additionally, 15 age/sex matched patients with stable RRMS who are not undergoing any change in treatment and are not currently on B-cell depleting therapies will be enrolled as control subjects.

ELIGIBILITY:
Inclusion Criteria:

For Ublituximab Group:

1. Ages 18-65
2. A diagnosis of relapsing MS (to include relapsing-remitting MS and active secondary progressive MS) according to 2017 Revised McDonald Criteria.
3. A recent referral for initiation of ublituximab for treatment of MS by the patient's treating physician.

For Comparison Group:

1. Ages 18 - 65
2. A diagnosis of relapsing-remitting MS according to 2017 Revised McDonald Criteria.
3. Currently on a stable dose of disease modifying treatment for MS with no plans for alternative therapy for the following year.

Exclusion Criteria:

For Ublituximab Group:

1. Known eye disease that may, in the opinion of the screening ophthalmologist, preclude proper analysis of data in this study. This includes, but is not limited to diabetic retinopathy, macular degeneration, and glaucoma.
2. Treatment with any B-cell depleting disease modifying therapy for MS (i.e. rituximab, ocrelizumab, ofatumumab, ublituximab, etc.) within the past 12 months.
3. History of life-threatening infusion reaction on ublituximab or prior anti-CD20 therapy
4. Any chronic or active infection that would preclude anti-CD20 therapy. This may include but is not limited to active hepatitis B virus (HBV) confirmed by positive results for Hepatitis B surface antigen (HBsAg) and anti-HBV tests, tuberculosis, and human immunodeficiency virus (HIV).
5. Receipt of any live of live-attenuated vaccines within 4 weeks prior to first ublituximab administration

For Comparison Group:

1. Known eye disease that may, in the opinion of the screening ophthalmologist, preclude proper analysis of data in this study. This includes, but is not limited to diabetic retinopathy, macular degeneration, and glaucoma.
2. Treatment with any B-cell depleting disease modifying therapy (i.e. rituximab, ocrelizumab, ofatumumab, ublituximab, etc.) within the past 12 months, or plans to initiate such a therapy in the following year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the effect of ublituximab on macular hyperreflective foci (HRF) in MS. | From enrollment until the last OCT at Months 6 and 12
  A change in the number of HRF seen on baseline compared to months 6 and 12 in the ublituximab grop compared to the comparison group
Evaluation of the effect of ublituximab on inner limiting membrane (ILM) macrophage-like cells (MLC). | From enrollment until the last OCT at Months 6 and 12
  A change in the number of MLCs seen from baseline to months 6 and 12 in the ublituximab group compared to the comparison group.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Harrison, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No